CLINICAL TRIAL: NCT02195154
Title: 18F-DTBZ PET and Multi-modal MRI in the Patients With Vascular Parkinsonism: Investigating the Correlation Between Cerebral Structural and Functional Changes, and Clinical Manifestation
Brief Title: 18F-DTBZ PET and Multi-modal MRI in the Patients With Vascular Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Wey-Yil Lin, Instructor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 101-4624A
Record Dates: First submitted 2014-02-27; First posted 2014-07-21 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Vascular Parkinsonism
Keywords: 18F-DTBZ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DTBZ for Vascular Parkinsonism (Experimental): This neuroimaging study includes the 18F-FP-(+)-DTBZ PET, MRI structure images, diffusion tensor imaging, susceptibility weighted imaging, resting state and gait-related imagery task functional MRI. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject group, each subject will have 3 visits in this study. Safety measurement for 18F-FP-(+)-DTBZ will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.
  Interventions: Drug: 18F-DTBZ

INTERVENTIONS:
Drug: 18F-DTBZ — During this study, subjects will receive a single i.v. administration of approximately 10 mCi 18F-FP-(+)-DTBZ immediately prior to imaging. The compound is labeled with fluorine 18F that decays by positron (β+) emission and has a half life of 109.7 min. The principal photons useful for diagnostic imaging are the 511 keV gamma photons, resulting from the interaction of the emitted positron with an electron.
  The proposed dose for this study is based on the phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG.

SUMMARY:
Forty patients with clinically diagnosed VP and 20 healthy subjects will be enrolled in the study. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria and each subject will have 3 visits in the study, as one screening visit, one imaging visit, and one safety evaluation visit.

DETAILED DESCRIPTION:
Study duration is expected to be completed in a period of 3 year. The study will enroll 40 patients with VP and 20 healthy subjects.

This neuroimaging study includes the 18F-FP-(+)-DTBZ PET, MRI structure images, diffusion tensor imaging, susceptibility weighted imaging, resting state and gait-related imagery task functional MRI. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject group, each subject will have 3 visits in this study. Safety measurement for 18F-FP-(+)-DTBZ will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Forty patients with a diagnosis of VP whom must: i. Male or female patients; age range 45~80 years old. ii. Written and dated informed consent by self or by legal representative, to be obtained before any of the study procedures.

iii. Patients should be fulfilled the diagnostic criteria of vascular parkinsonism (Appendix I).

2. Twenty healthy subjects whom must: i. Male or female patients; age range 45~80 years old. ii. Written and dated informed consent by self or by legal representative, to be obtained before any of the study procedures.

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.

   I. Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances.

   II. Current clinically significant cardiovascular disease. (cardiac surgery or myocardial infarction within the last 6 months; unstable angina; decompensated congestive heart failure; significant cardiac arrhythmia; congenital heart disease.)
3. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
4. History or presence of QTc prolongation.
5. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
6. History of repeated head injury, hydrocephalus, encephalitis or cerebral tumors.
7. History of neurotoxin exposure
8. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus or encephalomalacia, will be excluded. Cerebral vascular lesions are allowed for VP patients. Mild cortical atrophy will be allowed for all subjects.
9. Patients who have neurodegenerative diseases, such as spinocerellar atrophy (SCA), Wilson's disease, Parkinson's disease or Parkinson plus syndrome, are excluded.
10. General PET exclusion criteria.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
The difference of specific uptake ratio (SUR) of 18F-DTBZ between disease and control group | 3 years

SECONDARY OUTCOMES:
The correlation between parameters from different imaging modalities and the severity of motor symptoms or cognition in disease group. | 3 years
  The neuroimaging parameters include the SURs of 18F-DTBZ in each brain regions, diffusion indices in each brain regions, MARS score, and activated voxels in each brain regions from the gait-related imagery task functional MRI.

OTHER OUTCOMES:
The difference of diffusion indices obtained from DTI between disease and control group | 3 years
The difference of microbleed anatomical rating scale (MARS) score obtained from the SWI between disease and control group. | 3 years
The difference of functional connectivity maps associated with the seed region of interest (resting state functional MRI) between disease and control group. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memory Hospital, Taoyuan District, Taiwan